CLINICAL TRIAL: NCT02313155
Title: A Randomized Double Blind Parallel-Group Comparative Phase 1/2 Study to Evaluate the Safety and Immunogenicity of a Single Subcutaneous Injection of TAK-850 in Healthy Adult Subjects
Brief Title: Phase 1/2 Study of TAK-850 Subcutaneous Injection in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TAK-850/CPH-002; U1111-1164-1969 (Registry Identifier: UTN (WHO)); JapicCTI-142724 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-01

CONDITIONS: Influenza Infection
Keywords: Prevention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAK-850 0.5 mL (subcutaneous) (Experimental): Single subcutaneous injection of TAK-850
  Interventions: Drug: Subcutaneous injection of TAK-850
- TAK-850 0.5 mL (Intramuscular) (Experimental): Single intramuscular injection of TAK-850
  Interventions: Drug: Intramuscular injection of TAK-850

INTERVENTIONS:
Drug: Subcutaneous injection of TAK-850 — TAK-850 0.5 mL, Subcutaneous injection
  Arms: TAK-850 0.5 mL (subcutaneous)
Drug: Intramuscular injection of TAK-850 — TAK-850 0.5 mL, Intramuscular injection
  Arms: TAK-850 0.5 mL (Intramuscular)

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of a single subcutaneous injection of TAK-850 as compared to intramuscular injection of TAK-850 in healthy Japanese adults

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-850. This drug is being tested to evaluate the safety and immunogenicity of a single subcutaneous injection as compared to a single, intramuscular injection.

A total of 110 healthy participants (55 per group) will take part in this study.

Each participant will be randomly (like flipping a coin) assigned to receive one of the following :

* A single injection of TAK-850, subcutaneously , or
* A single injection of TAK-850, intramuscularly.

Participants will make up to 3 visits to the study site. Total duration of this study is 22 days.

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the investigator or subinvestigator, the participant is capable of understanding and complying with protocol requirements.

  2. The participant signs and dates a written, informed consent form prior to the initiation of any study procedures.

  3. The participant is a healthy Japanese adult male or female. 4. The participant is aged 20 to 49 years, inclusive, at the time of informed consent.

  5. The participant has a body mass index (BMI) between 18.5 and 25.0 kg/m^2, inclusive, at the time of eligibility evaluation.

  6. If the participant is a female of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study.

Exclusion Criteria:

* 1. The participant has received any investigational compound within 4 months prior to the injection of study vaccine.

  2. The participant has been vaccinated with seasonal influenza vaccine within 6 months prior to the injection of study vaccine.

  3. The participant has a history of influenza infection within 6 months prior to the injection of study vaccine.

  4. The participant is a study site employee, an immediate family member of such an employee, or in a dependent relationship with a study site employee who is involved in the conduct of this study (e.g., spouse, parent, child, sibling), or may consent under duress.

  5. The participant has uncontrolled, clinically significant manifestations of neurological, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, endocrine or other disorders, which may impact the ability of the participant to participate or potentially confound the study results.

  6. The participant has an oral temperature ≥37.5 °C prior to the injection of study vaccine on Day 1.

  7. The participant has any medically diagnosed or suspected immune deficient condition.

  8. The participant has an immune compromising condition or disease, or is currently undergoing a form of treatment or was undergoing a form of treatment that can be expected to influence immune response within 30 days prior to the injection of study vaccine. Such treatments include, but is not limited to, systemic or high dose inhaled corticosteroids (>800 mcg/day of beclomethasone dipropionate or equivalent; the use of inhaled and nasal steroids that do not exceed this level will be permitted), radiation treatment or other immunosuppressive or cytotoxic drugs.

  9. The participant has received antipyretics within 4 hours prior to the injection of study vaccine.

  10. The participant has a history of Guillain-Barré Syndrome, demyelinating disorders (including acute disseminated encephalomyelitis [ADEM] and multiple sclerosis) or convulsions.

  11. The participant has a functional or surgical asplenia. 12. The participant has a rash, other dermatologic conditions or tattoos which may interfere with the evaluation of injection site reaction as determined by the investigator.

  13. The participant has a history of, or is infected with the Hepatitis B Virus (HBsAgs), Hepatitis C Virus (HCV) or Human Immunodeficiency Virus (HIV).

  14. The participant has a known hypersensitivity to any component of TAK-850. 15. The participant has a history of severe allergic reactions or anaphylaxis. 16. The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the injection of study vaccine or is unwilling to agree to abstain from alcohol and drugs throughout the study.

  17. The participant has received any blood products (e.g. blood transfusion or immunoglobulin) within 90 days prior to the injection of study vaccine.

  18. The participant has received a live vaccine within 4 weeks (28 days) or an inactivated vaccine within 2 weeks (14 days) prior to the injection of study vaccine.

  19. If female, the participant is pregnant or lactating or intending to become pregnant before signing informed consent, during, or within 1 month after participating in this study; or intending to donate ova during such time period.

  20. The participant has donated whole blood ≥200 mL within 4 weeks (28 days), ≥400 mL within 12 weeks (84 days), ≥800 mL within 52 weeks (364 days), or blood components within 2 weeks (14 days) prior to the injection of study vaccine.

  21. The participant has abnormal laboratory values that suggest a clinically significant underlying disease at the assessment prior to the injection of study vaccine, or the participant has the following lab abnormalities: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) more than 3 times the upper limits of normal.

  22. In the opinion of the investigator or subinvestigator, the participant is unlikely to comply with protocol requirements or is considered ineligible for any other reason.

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2014-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior VP Clinical Science, Study Director — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Japan from 13-December-2014 to 22-January-2015.
Pre-assignment Details: Healthy adult participants were randomized to receive a single dose of 0.5 milliliter (mL) of TAK-850 in 1 of the 2 treatment groups: TAK-850 subcutaneous injection and TAK-850 intramuscular injection.
Groups:
- TAK-850 Subcutaneous Injection: TAK-850 0.5 mL (15 microgram [mcg] of hemagglutinin [HA] per strain), injection, subcutaneous, once on Day 1 in a treatment period of 22 days.
- TAK-850 Intramuscular Injection: TAK-850 0.5 mL (15 mcg of HA per strain), injection, intramuscular, once on Day 1 in a treatment period of 22 days.
Period: Overall Study
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Started | 55 | 55
Completed | 55 | 54
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set was defined as all participants who received vaccination with the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.1 (3.50) | 25.1 (4.08) | 24.6 (3.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 55
  Male | 28 | 27 | 55
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 165.9 (8.83) | 165.5 (8.67) | 165.7 (8.71)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 56.35 (7.325) | 58.19 (7.610) | 57.27 (7.492)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 20.41 (1.457) | 21.18 (1.561) | 20.79 (1.552)
Influenza Infection Within 1 Year [Number; unit: participants]
  Participant had influenza infection in 1 year (yr) | 0 | 1 | 1
  Participant didnot have influenza infection in 1yr | 55 | 54 | 109
Hemagglutination Inhibition (HI) (Egg-derived) - A/H1N1 at Day1 (Predose) Titer [Number; unit: participants] — Number of participants with values of HI antibody titer for A/H1N1 strain pre-dose at Day 1 were reported. Influenza A/Hemagglutinin Type 1 and Neuraminidase Type 1 (A/H1N1). Greater than or equal to (>=). Less than or equal to (<=).
  participants
    >=Minimum (Min) to <40 titer | 40 | 37 | 77
    >=40 to <=Maximum (Max) titer | 15 | 18 | 33
HI(Egg-derived) - A/H3N2 at Day1(Predose) Titer [Number; unit: participants] — Number of participants with values of HI antibody titer for A/H3N2 strain pre-dose at Day 1 were reported.
  participants
    >=Min to less than (<) 40 titer | 48 | 41 | 89
    >=40 to <=Max titer | 7 | 14 | 21
HI(Egg-derived) - Influenza B(B) at Day1(Predose) Titer [Number; unit: participants] — Number of participants with values of HI antibody titer for B strain pre-dose at Day 1 were reported.
  participants
    >=Min to < 40 titer | 25 | 25 | 50
    >=40 to <=Max titer | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Solicited Local and Systemic Adverse Events (AEs)
Description: Number of participants with local reactions (injection site pain, injection site redness, injection site swelling, injection site induration, injection site tenderness, and injection site ecchymosis) and systemic events (pyrexia, malaise, chills, fatigue, headache, sweaty, myalgia, arthralgia, nausea and vomiting) were reported using an electronic diary.
Time Frame: Up to 21 days (Day 22) after vaccination
Population: Safety analysis set was defined as all participants who received vaccination with the study drug.
Measure: Number; unit: participants
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Number analyzed (Participants) | 55 | 55
participants
  Injection site pain | 7 | 5
  Injection site redness | 4 | 0
  Injection site swelling | 4 | 0
  Injection site induration | 2 | 1
  Injection site tenderness | 29 | 26
  Injection site ecchymosis | 2 | 1
  Pyrexia | 2 | 2
  Malaise | 12 | 10
  Chills | 3 | 3
  Fatigue | 7 | 8
  Headache | 7 | 3
  Sweaty | 1 | 0
  Myalgia | 3 | 3
  Arthralgia | 4 | 3
  Nausea | 2 | 4

2. Primary Outcome: Number of Participants Who Experience at Least One Treatment Emergent Adverse Event (TEAE)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Up to 21 days (Day 22) after vaccination
Population: Safety analysis set was defined as all participants who received vaccination with the study drug.
Measure: Number; unit: participants
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Number analyzed (Participants) | 55 | 55
participants | 34 | 32

3. Primary Outcome: Percentage of Participants With Seroprotection in Hemagglutination Inhibition (HI) Antibody Titer (Egg-derived Antigen) of >=40.
Description: Seroprotection rate as measured by HI antibody titer (egg-derived antigen) was defined as percentage of participants with the HI antibody titer of >=40 for each of the three influenza virus strains (A/H1N1 strain, A/H3N2 strain, and B strain).
Time Frame: Day 22 (21 days after vaccination)
Population: Full analysis set was defined as participants who were randomized and received vaccination with the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Number analyzed (Participants) | 55 | 54
percentage of participants
  A/H1N1 strain | 80.0 [67.027 to 89.570] | 88.9 [77.369 to 95.812]
  A/H3N2 strain | 49.1 [35.354 to 62.929] | 70.4 [56.391 to 82.022]
  B strain | 87.3 [75.520 to 94.726] | 90.7 [79.700 to 96.925]

4. Primary Outcome: Percentage of Participants With Seroconversion in Hemagglutination Inhibition (HI) Antibody Titer (Egg-Derived Antigen)
Description: Seroconversion rate as measured by the HI antibody titer (egg-derived antigen) was defined as percentage of participants achieving a minimal 4-fold increase from the baseline HI antibody titer (baseline >=10) or achieving an HI antibody titer of >=40 (baseline <10) for each of the three influenza virus strains (A/H1N1 strain, A/H3N2 strain, and B strain).
Time Frame: Day 22 (21 days after vaccination)
Population: Full analysis set was defined as participants who were randomized and received vaccination with the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Number analyzed (Participants) | 55 | 54
percentage of participants
  A/H1N1 strain | 58.2 [44.106 to 71.345] | 64.8 [50.624 to 77.319]
  A/H3N2 strain | 34.5 [22.237 to 48.581] | 50.0 [36.081 to 63.919]
  B strain | 34.5 [22.237 to 48.581] | 46.3 [32.622 to 60.391]
Statistical Analysis 1: Comparison: TAK-850 Subcutaneous Injection vs TAK-850 Intramuscular Injection; A/H1N1 Strain; Test type: Superiority or Other; Difference = -6.6, 95% CI 2-sided [-24.858 to 11.592] — Seroconversion rate difference between treatment groups was obtained by subtracting the value of TAK-850 I.M. from TAK-850 S.C
Statistical Analysis 2: Comparison: TAK-850 Subcutaneous Injection vs TAK-850 Intramuscular Injection; A/H3N2 Strain; Test type: Superiority or Other; Difference = -15.5, 95% CI 2-sided [-33.779 to 2.870] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: TAK-850 Subcutaneous Injection vs TAK-850 Intramuscular Injection; B Strain; Test type: Superiority or Other; Difference = -11.8, 95% CI 2-sided [-30.048 to 6.547] — [estimate comment as in outcome 4, analysis 1]

5. Primary Outcome: Geometric Mean Fold Increase (GMFI) in HI Antibody Titer (Egg-derived Antigen) From Pre-vaccination to 21 Days After Vaccination
Description: GMFI in HI antibody titer (egg-derived antigen) as compared to pre-vaccination was evaluated for each of the three influenza virus strains (A/H1N1 strain, A/H3N2 strain, and B strain). Geometric mean and CI were calculated for GMFIs.
Time Frame: Pre-vaccination, 21 Days After vaccination (Day 22)
Population: Full analysis set was defined as participants who were randomized and received vaccination with the study drug.
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Number analyzed (Participants) | 55 | 54
fold increase
  A/H1N1 strain | 10.23 [5.939 to 17.616] | 15.54 [8.922 to 27.082]
  A/H3N2 strain | 3.01 [2.003 to 4.530] | 4.40 [2.898 to 6.693]
  B strain | 3.70 [2.632 to 5.192] | 4.13 [2.886 to 5.912]

6. Secondary Outcome: Number of Participants Reporting Clinically Significant Change From Baseline in Laboratory Values
Description: Laboratory values included hematology, biochemistry and urinalysis tests.
Time Frame: Baseline,up to 21 Days after drug administration (Day 22)
Population: Safety analysis set was defined as all participants who received vaccination with the study drug.
Measure: Number; unit: participants
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Number analyzed (Participants) | 55 | 55
participants | 2 | 1

7. Secondary Outcome: Change From Baseline in Blood Pressure
Description: Change from baseline in systolic and diastolic blood pressure was reported
Time Frame: Baseline, Day 22
Population: Safety analysis set was defined as all participants who received vaccination with the study drug.
Measure: Mean (Standard Deviation); unit: millimeter mercury (mmHg)
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Number analyzed (Participants) | 55 | 55
millimeter mercury (mmHg)
  Systolic Blood Pressure: Baseline | 109.3 (11.36) | 112.2 (10.93)
  Systolic Blood Pressure: Change at Day 22 | -0.7 (9.78) | -0.9 (9.94)
  Diastolic Blood Pressure: Baseline | 63.8 (7.50) | 66.3 (8.57)
  Diastolic Blood Pressure: Change at Day 22 | 0.4 (7.47) | 0.4 (6.89)

8. Secondary Outcome: Change From Baseline in Pulse
Description: Change from baseline in pulse was reported.
Time Frame: Baseline, Day 22
Population: Safety analysis set was defined as all participants who received vaccination with the study drug.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Number analyzed (Participants) | 55 | 55
beats per minute
  Pulse: Baseline | 72.9 (11.69) | 72.9 (10.34)
  Pulse: Change at Day 22 | -2.3 (11.35) | -2.0 (8.51)

9. Secondary Outcome: Change From Baseline in Body Temperature
Description: Change from baseline in body temperature (oral) was reported.
Time Frame: Baseline, Day 22
Population: Safety analysis set was defined as all participants who received vaccination with the study drug.
Measure: Mean (Standard Deviation); unit: degree celsius
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Number analyzed (Participants) | 55 | 55
degree celsius
  Temperature: Baseline | 36.71 (0.305) | 36.72 (0.311)
  Temperature: Change at Day 22 | -0.21 (0.357) | -0.20 (0.388)

10. Secondary Outcome: Geometric Mean Titer (GMT) in HI Antibody Titer (Egg-derived Antigen)
Description: GMT in HI antibody titer (egg-derived antigen) for each of the three influenza virus strains (A/H1N1 strain, A/H3N2 strain, and B strain) was computed along with 95% CI.
Time Frame: Day 22 (21 days after vaccination)
Population: Full analysis set was defined as participants who were randomized and received vaccination with the study drug.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Number analyzed (Participants) | 55 | 54
titer
  A/H1N1 strain | 143.30 [87.531 to 234.589] | 237.43 [156.037 to 361.284]
  A/H3N2 strain | 21.91 [14.256 to 33.683] | 51.21 [32.446 to 80.835]
  B strain | 82.56 [59.943 to 113.715] | 107.13 [78.013 to 147.122]

11. Secondary Outcome: Percentage of Participants With Seroprotection in SRH Antibody Titer (Egg-derived Antigen) of >=25 mm^2
Description: Seroprotection rate as measured by SRH antibody titer (egg-derived antigen) was defined as percentage of participants with an SRH antibody titer of >=25 mm^2 for each of the three influenza virus strains (A/H1N1 strain, A/H3N2 strain, and B strain).
Time Frame: Day 22 (21 days after vaccination)
Population: Full analysis set was defined as participants who were randomized and received vaccination with the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Number analyzed (Participants) | 55 | 54
percentage of participants
  A/H1N1 strain | 100.0 [93.513 to 100.000] | 100.0 [93.397 to 100.000]
  A/H3N2 strain | 67.3 [53.293 to 79.319] | 75.9 [62.359 to 86.514]
  B strain | 100.0 [93.513 to 100.000] | 100.0 [93.397 to 100.000]

12. Secondary Outcome: Percentage of Participants With Seroconversion in SRH Antibody Titer (Egg-Derived Antigen)
Description: Seroconversion rate as measured by the SRH antibody titer (egg-derived antigen) was defined as percentage of participants achieving a minimal 50% increase from the baseline SRH antibody titer (baseline >4 mm^2) or achieving an SRH antibody titer of >=25 mm^2 (baseline <=4 mm^2) for each of the three influenza virus strains (A/H1N1 strain, A/H3N2 strain, and B strain).
Time Frame: Day 22 (21 days after vaccination)
Population: Full analysis set was defined as participants who were randomized and received vaccination with the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Number analyzed (Participants) | 55 | 54
percentage of participants
  A/H1N1 strain | 58.2 [44.106 to 71.345] | 61.1 [46.879 to 74.080]
  A/H3N2 strain | 41.8 [28.655 to 55.894] | 51.9 [37.837 to 65.657]
  B strain | 38.2 [25.409 to 52.274] | 46.3 [32.622 to 60.391]

13. Secondary Outcome: GMFI in SRH Antibody Titer (Egg-derived Antigen) From Pre-vaccination to 21 Days After Vaccination
Description: GMFI in SRH antibody titer (egg-derived antigen) as compared to baseline pre-vaccination was evaluated for each of the three influenza virus strains (A/H1N1 strain, A/H3N2 strain, and B strain). Geometric mean and CI were calculated for GMFIs.
Time Frame: Pre-vaccination, 21 Days after vaccination (Day 22)
Population: Full analysis set was defined as participants who were randomized and received vaccination with the study drug.
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Number analyzed (Participants) | 55 | 54
fold increase
  A/H1N1 strain | 2.5435 [1.98252 to 3.26315] | 2.4169 [1.87743 to 3.11144]
  A/H3N2 strain | 1.7666 [1.46398 to 2.13181] | 2.3687 [1.86326 to 3.01124]
  B strain | 1.5867 [1.37637 to 1.82926] | 1.6380 [1.42438 to 1.88370]

14. Secondary Outcome: GMT in SRH Antibody Titer (Egg-derived Antigen)
Description: GMT in SRH antibody titer (egg-derived antigen) for each of the three influenza virus strains (A/H1N1 strain, A/H3N2 strain, and B strain) was computed along with 95% CI.
Time Frame: Day 22 (21 days after vaccination)
Population: Full analysis set was defined as participants who were randomized and received vaccination with the study drug.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Number analyzed (Participants) | 55 | 54
titer
  A/H1N1 strain | 75.5840 [69.35268 to 82.37530] | 82.4482 [77.42068 to 87.80227]
  A/H3N2 strain | 28.9569 [23.40813 to 35.82096] | 34.0601 [27.64669 to 41.96127]
  B strain | 70.5747 [67.07223 to 74.26000] | 73.2954 [69.23834 to 77.59029]

15. Secondary Outcome: Percentage of Participants With Seroprotection in HI Antibody Titer (Cell Derived Antigen) of >=40
Description: Seroprotection rate as measured by HI antibody titer (vero antigen, live-vero antigen, and madin-darby canine kidney [MDCK] antigen) was defined as percentage of participants with an HI antibody titer of >=40 for each of the three influenza virus strains (A/H1N1 strain, A/H3N2 strain, and B strain).
Time Frame: Day 22 (21 days after vaccination)
Population: Full analysis set was defined as participants who were randomized and received vaccination with the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Number analyzed (Participants) | 55 | 54
percentage of participants
  Vero antigen: A/H1N1 strain | 41.8 [28.655 to 55.894] | 46.3 [32.622 to 60.391]
  Vero antigen: A/H3N2 strain | 41.8 [28.655 to 55.894] | 55.6 [41.400 to 69.080]
  Vero antigen: B strain | 60.0 [45.907 to 72.977] | 72.2 [58.356 to 83.545]
  Live-Vero antigen: A/H1N1 strain | 92.7 [82.413 to 97.983] | 98.1 [90.108 to 99.953]
  Live-Vero antigen: A/H3N2 strain | 96.4 [87.474 to 99.557] | 96.3 [87.253 to 99.548]
  Live-Vero antigen: B strain | 96.4 [87.474 to 99.557] | 94.4 [84.611 to 98.839]
  MDCK antigen: A/H1N1 strain | 90.9 [80.046 to 96.982] | 98.1 [90.108 to 99.953]
  MDCK antigen: A/H3N2 strain | 92.7 [82.413 to 97.983] | 92.6 [82.107 to 97.945]
  MDCK antigen: B strain | 98.2 [90.281 to 99.954] | 94.4 [84.611 to 98.839]

16. Secondary Outcome: Percentage of Participants With Seroconversion in HI Antibody Titer (Cell Derived Antigen)
Description: Seroconversion rate as measured by the HI antibody titer (vero antigen, live-vero antigen, and madin-darby canine kidney [MDCK] antigen) was defined as percentage of participants achieving a minimal 4-fold increase from the baseline HI antibody titer (baseline >=10) or achieving an HI antibody titer of >=40 (baseline HI <10) for each of the three influenza virus strains (A/H1N1 strain, A/H3N2 strain, and B strain).
Time Frame: Day 22 (21 days after vaccination)
Population: Full analysis set was defined as participants who were randomized and received vaccination with the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Number analyzed (Participants) | 55 | 54
percentage of participants
  Vero antigen: A/H1N1 strain | 41.8 [28.655 to 55.894] | 42.6 [29.235 to 56.792]
  Vero antigen: A/H3N2 strain | 36.4 [23.814 to 50.437] | 50.0 [36.081 to 63.919]
  Vero antigen: B strain | 34.5 [22.237 to 48.581] | 48.1 [34.343 to 62.163]
  Live-Vero antigen: A/H1N1 strain | 54.5 [40.554 to 68.030] | 70.4 [56.391 to 82.022]
  Live-Vero antigen: A/H3N2 strain | 40.0 [27.023 to 54.093] | 50.0 [36.081 to 63.919]
  Live-Vero antigen: B strain | 32.7 [20.681 to 46.707] | 38.9 [25.920 to 53.121]
  MDCK antigen: A/H1N1 strain | 45.5 [31.970 to 59.446] | 61.1 [46.879 to 74.080]
  MDCK antigen: A/H3N2 strain | 47.3 [33.653 to 61.196] | 57.4 [43.208 to 70.765]
  MDCK antigen: B strain | 32.7 [20.681 to 46.707] | 33.3 [21.092 to 47.474]

17. Secondary Outcome: GMFI in HI Antibody Titer (Cell Derived Antigen) From Pre-vaccination to 21 Days After Vaccination
Description: GMFI in HI antibody titer (vero antigen, live-vero antigen, and madin-darby canine kidney [MDCK] antigen) as compared to pre-vaccination was evaluated for each of the three influenza virus strains (A/H1N1 strain, A/H3N2 strain, and B strain). Geometric mean and CI were calculated for GMFIs.
Time Frame: Pre-vaccination, 21 Days After vaccination (Day 22)
Population: Full analysis set was defined as participants who were randomized and received vaccination with the study drug.
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Number analyzed (Participants) | 55 | 54
fold increase
  Vero antigen: A/H1N1 strain | 3.10 [2.101 to 4.570] | 3.51 [2.311 to 5.321]
  Vero antigen: A/H3N2 strain | 2.66 [1.872 to 3.791] | 4.17 [2.792 to 6.228]
  Vero antigen: B strain | 2.84 [2.069 to 3.891] | 3.74 [2.666 to 5.246]
  Live-Vero antigen: A/H1N1 strain | 7.95 [5.012 to 12.609] | 12.70 [7.823 to 20.614]
  Live-Vero antigen: A/H3N2 strain | 3.95 [2.684 to 5.812] | 5.88 [3.835 to 9.013]
  Live-Vero antigen: B strain | 3.19 [2.336 to 4.351] | 3.66 [2.717 to 4.920]
  MDCK antigen: A/H1N1 strain | 5.95 [3.767 to 9.396] | 9.12 [5.740 to 14.505]
  MDCK antigen: A/H3N2 strain | 5.52 [3.609 to 8.431] | 8.10 [4.931 to 13.315]
  MDCK antigen: B strain | 3.67 [2.516 to 5.364] | 3.45 [2.483 to 4.796]

18. Secondary Outcome: GMT in HI Antibody Titer (Cell Derived Antigen)
Description: GMT in HI antibody titer (vero antigen, live-vero antigen, and madin-darby canine kidney [MDCK] antigen) for each of the three influenza virus strains (A/H1N1 strain, A/H3N2 strain, and B strain) was computed along with 95% CI.
Time Frame: Day 22 (21 days after vaccination)
Population: Full analysis set was defined as participants who were randomized and received vaccination with the study drug.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Number analyzed (Participants) | 55 | 54
titer
  Vero antigen: A/H1N1 strain | 17.52 [11.513 to 26.666] | 20.72 [13.374 to 32.096]
  Vero antigen: A/H3N2 strain | 17.63 [11.714 to 26.540] | 32.05 [20.018 to 51.327]
  Vero antigen: B strain | 27.24 [18.672 to 39.731] | 37.40 [26.335 to 53.102]
  Live-Vero antigen: A/H1N1 strain | 276.83 [192.610 to 397.866] | 424.41 [317.572 to 567.203]
  Live-Vero antigen: A/H3N2 strain | 208.48 [154.101 to 282.045] | 320.00 [225.694 to 453.713]
  Live-Vero antigen: B strain | 139.29 [113.528 to 170.887] | 168.43 [125.641 to 225.795]
  MDCK antigen: A/H1N1 strain | 257.47 [171.653 to 386.187] | 381.77 [289.028 to 504.274]
  MDCK antigen: A/H3N2 strain | 187.89 [132.545 to 266.336] | 309.89 [208.367 to 460.871]
  MDCK antigen: B strain | 187.89 [151.967 to 232.298] | 210.85 [155.714 to 285.513]

19. Secondary Outcome: Percentage of Participants With Seroprotection in SRH Antibody Titer (Cell Derived Antigen) of >=25 mm^2
Description: Seroprotection rate as measured by SRH antibody titer (vero antigen, live-vero antigen, and madin-darby canine kidney [MDCK] antigen) was defined as percentage of participants with a SRH antibody titer of >=25 mm^2 for each of the three influenza virus strains (A/H1N1 strain, A/H3N2 strain, and B strain).
Time Frame: Day 22 (21 days after vaccination)
Population: Full analysis set was defined as participants who were randomized and received vaccination with the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Number analyzed (Participants) | 55 | 54
percentage of participants
  Vero antigen: A/H1N1 strain | 76.4 [62.980 to 86.772] | 70.4 [56.391 to 82.022]
  Vero antigen: A/H3N2 strain | 98.2 [90.281 to 99.954] | 100 [93.397 to 100.000]
  Vero antigen: B strain | 98.2 [90.281 to 99.954] | 100 [93.397 to 100.000]
  Live-Vero antigen: A/H1N1 strain | 98.2 [90.281 to 99.954] | 100 [93.397 to 100.000]
  Live-Vero antigen: A/H3N2 strain | 100 [93.513 to 100.000] | 100 [93.397 to 100.000]
  Live-Vero antigen: B strain | 100 [93.513 to 100.000] | 100 [93.397 to 100.000]
  MDCK antigen: A/H1N1 strain | 89.1 [77.753 to 95.890] | 94.4 [84.611 to 98.839]
  MDCK antigen: A/H3N2 strain | 94.5 [84.877 to 98.861] | 98.1 [90.108 to 99.953]
  MDCK antigen: B strain | 100 [93.513 to 100.000] | 100 [93.397 to 100.000]

20. Secondary Outcome: Percentage of Participants With Seroconversion in SRH Antibody Titer (Cell Derived Antigen)
Description: Seroconversion rate as measured by the SRH antibody titer (vero antigen, live-vero antigen, and madin-darby canine kidney [MDCK] antigen) was defined as percentage of participants achieving a minimal 50% increase from the baseline SRH antibody titer (baseline >4 mm^2) or achieving an SRH antibody titer of >=25 mm^2 (baseline <=4 mm^2) for each of the three influenza virus strains (A/H1N1 strain, A/H3N2 strain, and B strain).
Time Frame: Day 22 (21 days after vaccination)
Population: Full analysis set was defined as participants who were randomized and received vaccination with the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Number analyzed (Participants) | 55 | 54
percentage of participants
  Vero antigen: A/H1N1 strain | 61.8 [47.726 to 74.591] | 63.0 [48.742 to 75.709]
  Vero antigen: A/H3N2 strain | 72.7 [59.038 to 83.862] | 77.8 [64.400 to 87.956]
  Vero antigen: B strain | 45.5 [31.970 to 59.446] | 44.4 [30.920 to 58.600]
  Live-Vero antigen: A/H1N1 strain | 50.9 [37.071 to 64.646] | 46.3 [32.622 to 60.391]
  Live-Vero antigen: A/H3N2 strain | 38.2 [25.409 to 52.274] | 44.4 [30.920 to 58.600]
  Live-Vero antigen: B strain | 34.5 [22.237 to 48.581] | 48.1 [34.343 to 62.163]
  MDCK antigen: A/H1N1 strain | 58.2 [44.106 to 71.345] | 61.1 [46.879 to 74.080]
  MDCK antigen: A/H3N2 strain | 47.3 [33.653 to 61.196] | 55.6 [41.400 to 69.080]
  MDCK antigen: B strain | 34.5 [22.237 to 48.581] | 38.9 [25.920 to 53.121]

21. Secondary Outcome: GMFI in SRH Antibody Titer (Cell Derived Antigen) From Pre-vaccination to 21 Days After Vaccination
Description: GMFI in SRH antibody titer (vero antigen, live-vero antigen, and madin-darby canine kidney [MDCK] antigen) as compared to pre-vaccination was evaluated for each of the three influenza virus strains (A/H1N1 strain, A/H3N2 strain, and B strain). Geometric mean and CI were calculated for GMFIs.
Time Frame: Pre-vaccination, 21 Days After vaccination (Day 22)
Population: Full analysis set was defined as participants who were randomized and received vaccination with the study drug.
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Number analyzed (Participants) | 55 | 54
fold increase
  Vero antigen: A/H1N1 strain | 2.8410 [2.27071 to 3.55446] | 3.4599 [2.68443 to 4.45933]
  Vero antigen: A/H3N2 strain | 2.2144 [1.90391 to 2.57562] | 2.4938 [2.09701 to 2.96573]
  Vero antigen: B strain | 1.7421 [1.49521 to 2.02974] | 1.7632 [1.51939 to 2.04622]
  Live-Vero antigen: A/H1N1 strain | 2.4134 [1.77374 to 3.28374] | 2.4059 [1.77115 to 3.26809]
  Live-Vero antigen: A/H3N2 strain | 2.0173 [1.53910 to 2.64419] | 2.2430 [1.69452 to 2.96898]
  Live-Vero antigen: B strain | 1.7655 [1.42885 to 2.18152] | 1.8173 [1.49254 to 2.21278]
  MDCK antigen: A/H1N1 strain | 2.6215 [2.03478 to 3.37729] | 3.1694 [2.38685 to 4.20840]
  MDCK antigen: A/H3N2 strain | 2.6078 [1.98732 to 3.42193] | 2.8178 [2.10367 to 3.77438]
  MDCK antigen: B strain | 1.6128 [1.37610 to 1.89014] | 1.5651 [1.35121 to 1.81284]

22. Secondary Outcome: GMT in SRH Antibody Titer (Cell Derived Antigen)
Description: GMT in SRH antibody titer (vero antigen, live-vero antigen, and madin-darby canine kidney [MDCK] antigen) for each of the three influenza virus strains (A/H1N1 strain, A/H3N2 strain, and B strain) was computed along with 95% CI.
Time Frame: Day 22 (21 days after vaccination)
Population: Full analysis set was defined as participants who were randomized and received vaccination with the study drug.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Number analyzed (Participants) | 55 | 54
titer
  Vero antigen: A/H1N1 strain | 29.2669 [24.46183 to 35.01576] | 33.3318 [27.94941 to 39.75064]
  Vero antigen: A/H3N2 strain | 53.3488 [48.65362 to 58.49703] | 57.3376 [52.02305 to 63.19507]
  Vero antigen: B strain | 51.4941 [47.87718 to 55.38425] | 54.3183 [50.64237 to 58.26095]
  Live-Vero antigen: A/H1N1 strain | 77.3268 [68.22339 to 87.64491] | 87.2200 [82.62689 to 92.06834]
  Live-Vero antigen: A/H3N2 strain | 75.9017 [70.70835 to 81.47657] | 79.7297 [73.82638 to 86.10500]
  Live-Vero antigen: B strain | 77.4468 [73.26937 to 81.86249] | 82.3667 [78.50179 to 86.42200]
  MDCK antigen: A/H1N1 strain | 43.3793 [36.13208 to 52.08009] | 51.8747 [46.86724 to 57.41712]
  MDCK antigen: A/H3N2 strain | 52.7714 [45.49007 to 61.21810] | 60.2234 [52.03699 to 69.69772]
  MDCK antigen: B strain | 83.9627 [79.99444 to 88.12783] | 87.5052 [83.09898 to 92.14495]

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs will be defined as any AEs, regardless of relationship to study drug, that occur or worsen after the dose of study drug and no more than 21 days after the study drug administration (up to Day 22).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-850 Subcutaneous Injection | TAK-850 Intramuscular Injection
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 34/55 | 32/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-850 Subcutaneous Injection (N=55) | TAK-850 Intramuscular Injection (N=55)
Nausea (Gastrointestinal disorders) | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Injection site pain (General disorders) | 29 | 28
Malaise (General disorders) | 12 | 10
Fatigue (General disorders) | 7 | 8
Injection site pruritus (General disorders) | 8 | 2
Chills (General disorders) | 3 | 3
Injection site erythema (General disorders) | 4 | 0
Injection site swelling (General disorders) | 4 | 0
Pyrexia (General disorders) | 2 | 2
Injection site haemorrhage (General disorders) | 2 | 1
Injection site induration (General disorders) | 2 | 1
Injection site warmth (General disorders) | 1 | 1
Feeling hot (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 4 | 2
Gastroenteritis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Headache (Nervous system disorders) | 7 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.